CLINICAL TRIAL: NCT06536777
Title: Effects of Ballistic Six Exercises With and Without Blood Flow Restriction on Agility, Strength and Functional Ability in Cricket Players
Brief Title: Effects of Ballistic Six Exercises With and Without Blood Flow Restriction in Cricket Players
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR & AHS/23/0468
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Plyometric Exercise; Blood Flow Restriction Training
Keywords: Plyometric training; Blood flow restriction
MeSH Terms: interventions — Plyometric Exercise; Blood Flow Restriction Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Clinical Trial
Who Masked: Outcomes Assessor
Masking Description: The assessor who will take the readings is blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plyometric Training (Active Comparator): Ballistic six exercises (Elastic ER, Elastic 90/90 ER, Overhead throw, 90/90 flexion ER Decel Throw, 90/90 Abduction ER Decel Throw, Internal Rotation). Ballistic Six plyometric training, done 2 days a week for 8 weeks, was given to the bowlers for rotator cuff muscles of their dominant shoulders. Exercises were performed using 3 sets of 10-20 repetitions, with 30 s of rest between each set. The progression of the training protocol. The equipment utilized in the Ballistic Six exercises included medicine balls (2-lb for single arm exercises and 6-lb for the 2-handed exercises). Subjects continued their strength and conditioning activities in off-season along with the Ballistic Six exercises. Following 8 weeks of training, post-readings for the bowling velocity, identical to that described in the pretesting protocol, were obtained and documented.
  Interventions: Other: Plyometric Exercises
- Plyometric Training with Blood Flow Resistance Training (Experimental): Experiment group received Ballistic six exercises with Blood Flow Restriction (BFR) training. Regularly monitor and supervise the training sessions. BFR training is a method that mimics the effects of high intensity training by combining low intensity exercise with blood flow obstruction. A pneumatic cuff, often known as a tourniquet, is applied proximally to the muscle that is being trained. It can be used on the lower or upper extremity. The next step is to inflate the cuff to a certain pressure in order to achieve both total and partial venous blockage. The patient is then instructed to conduct resistance exercises with high repetitions (15-30) and short rest periods (30 sec) at a low intensity of 20-30% of 1 repetition maximum (1RM).
  Interventions: Other: Plyometric Exercises; Other: Blood Flow Restriction Training

INTERVENTIONS:
Other: Plyometric Exercises — This include Plyometric Training for 8 weeks
Other: Blood Flow Restriction Training — This include Blood Flow Restriction Training for 8 weeks
  Arms: Plyometric Training with Blood Flow Resistance Training

SUMMARY:
Cricket is not only a widely played team sport, but it also involves intricate skills that are honed over time, especially in bowling. One of the key concerns for bowlers is the risk of developing shoulder injuries due to imbalances between the agonist and antagonist muscle groups. To address this, the Ballistic Six program focuses on functional exercises that replicate the movements and forces involved in the overhead throwing motion, helping to enhance strength, power, proprioception, kinesthesia, and endurance in the rotator cuff muscles. By incorporating plyometric training in a ballistic, high-velocity manner, the program aims to take advantage of the stretch reflex and reduce the amortization phase of the stretch shortening cycle. Additionally, blood flow restriction (BFR) training has shown promising results in promoting muscle growth and strength. By applying a tourniquet to the arm during intra-set rests, BFR induces muscle hypoxia while restricting venous return, leading to increased lean mass, isometric strength, and muscular endurance in the shoulder and arm. These training methods can contribute to the overall performance and injury prevention of medium pace cricket bowlers.

DETAILED DESCRIPTION:
In addition to being a popular team activity, cricket requires complex abilities that are developed through time, particularly in bowling. The possibility of shoulder injuries resulting from imbalances between the agonist and antagonist muscle groups is one of the main worries for bowlers. The Ballistic Six program aims to improve the rotator cuff muscles' strength, power, proprioception, kinesthesia, and endurance by using functional exercises that mimic the motions and pressures involved in the overhead throwing action. The program's goal is to minimize the stretch shortening cycle's amortization phase and maximize the stretch reflex by combining plyometric training in a ballistic, high-velocity way. Furthermore, training with blood flow restriction (BFR) has demonstrated encouraging outcomes in enhancing muscle mass and power. Lean mass, isometric strength, and muscular endurance in the shoulder and arm are enhanced by BFR, which produces muscle hypoxia while limiting venous return by placing a tourniquet to the arm during intra-set rests. Medium-pace cricket bowlers can benefit from these training techniques in terms of both overall performance and injury prevention.

To maintain fairness in this Randomized Controlled Trial, volunteers will be chosen at random. The 18-25-year-old cricket players will be split into two groups: an experimental group and a control group. Ballistic Six upper extremity plyometric training will be administered to the control group, while Ballistic Six training combined with blood flow restriction treatment will be administered to the experimental group. The course of therapy will last for eight weeks, with monthly progress reports. There will be three weekly recovery sessions, each lasting 20 to 30 minutes. Tests such as the Kerlan Jobe Orthopedic Clinic (KJOC) Shoulder and Elbow Score, the Closed Kinetic Chain Upper Extremity Stability Test, and the Seated Medicine Ball Throw Test will be used to assess patients both at the start and finish of their therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male players
* Age 18-25 years
* Active recreational players
* Minimum score on Kerlan-Jobe Orthopedic Clinic (KJOC) Shoulder and Elbow Score questionnaire should be above 60.
* In Closed kinetic chain upper extremity stability test rest interval should be from 40-45 seconds.
* Athletes playing cricket with minimum 1 year experience

Exclusion Criteria:

* Players not actively involved in training and competition
* History of systemic disease
* Prior surgery history
* Ligamentous and GHJ injury
* Bone deformity
* Fractures of upper limb
* Vestibular and visual disorder
* Pre-existing shoulder pathologies or injuries

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 32 (Estimated)
Dates: Start 2024-06-25 (Actual); Primary Completion 2024-09-25 (Estimated); Study Completion 2024-09-25 (Estimated)

PRIMARY OUTCOMES:
Agility | 0 week, 8 week
  Will be measured by Closed Kinetic Chain Upper Extremity Stability (CKCUES) Test
Strength | 0 week, 8 week
  Will be measured by Seated medicine ball throw test
Functional Ability | 0 week, 8 week
  Will be measured by Kerlan-Jobe Orthopaedic Clinic (KJOC) Shoulder and Elbow Score

CONTACTS AND LOCATIONS:
Overall Officials: Mahnoor Majid, DPT, Principal Investigator — Riphah International University
Locations (1):
- Dring Stadium, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ali K, Gupta S, Hussain ME, Alzhrani M, Manzar MD, Khan M, Alghadir AH. Effect of plyometric versus complex training on core strength, lower limb, and upper limb power in male cricketers: a randomized controlled trial. BMC Sports Sci Med Rehabil. 2023 Nov 27;15(1):160. doi: 10.1186/s13102-023-00771-8. PMID 38008712
- [Background] Singla D, Hussain ME. Adaptations of the Upper Body to Plyometric Training in Cricket Players of Different Age Groups. J Sport Rehabil. 2019 Oct 18;29(6):697-706. doi: 10.1123/jsr.2018-0469. Print 2020 Aug 1. PMID 31141445
- [Background] Maker R, Taliep MS. The effects of a four weeks combined resistance training programme on cricket bowling velocity. S Afr J Sports Med. 2021 Jun 10;33(1):v33i1a9002. doi: 10.17159/2078-516X/2021/v33i1a9002. eCollection 2021. PMID 36816886
- [Background] Grgic J, Schoenfeld BJ, Mikulic P. Effects of plyometric vs. resistance training on skeletal muscle hypertrophy: A review. J Sport Health Sci. 2021 Sep;10(5):530-536. doi: 10.1016/j.jshs.2020.06.010. Epub 2020 Jun 21. PMID 32579911
- [Background] Ramirez-Campillo R, Garcia-Hermoso A, Moran J, Chaabene H, Negra Y, Scanlan AT. The effects of plyometric jump training on physical fitness attributes in basketball players: A meta-analysis. J Sport Health Sci. 2022 Nov;11(6):656-670. doi: 10.1016/j.jshs.2020.12.005. Epub 2020 Dec 24. PMID 33359798
- [Background] Erickson LN, Lucas KCH, Davis KA, Jacobs CA, Thompson KL, Hardy PA, Andersen AH, Fry CS, Noehren BW. Effect of Blood Flow Restriction Training on Quadriceps Muscle Strength, Morphology, Physiology, and Knee Biomechanics Before and After Anterior Cruciate Ligament Reconstruction: Protocol for a Randomized Clinical Trial. Phys Ther. 2019 Aug 1;99(8):1010-1019. doi: 10.1093/ptj/pzz062. PMID 30951598
- [Background] Pignanelli C, Christiansen D, Burr JF. Blood flow restriction training and the high-performance athlete: science to application. J Appl Physiol (1985). 2021 Apr 1;130(4):1163-1170. doi: 10.1152/japplphysiol.00982.2020. Epub 2021 Feb 18. PMID 33600282
- [Background] Wortman RJ, Brown SM, Savage-Elliott I, Finley ZJ, Mulcahey MK. Blood Flow Restriction Training for Athletes: A Systematic Review. Am J Sports Med. 2021 Jun;49(7):1938-1944. doi: 10.1177/0363546520964454. Epub 2020 Nov 16. PMID 33196300
- [Background] Hwang PS, Willoughby DS. Mechanisms Behind Blood Flow-Restricted Training and its Effect Toward Muscle Growth. J Strength Cond Res. 2019 Jul;33 Suppl 1:S167-S179. doi: 10.1519/JSC.0000000000002384. PMID 30011262
- [Background] Lambert B, Hedt C, Daum J, Taft C, Chaliki K, Epner E, McCulloch P. Blood Flow Restriction Training for the Shoulder: A Case for Proximal Benefit. Am J Sports Med. 2021 Aug;49(10):2716-2728. doi: 10.1177/03635465211017524. Epub 2021 Jun 10. PMID 34110960